CLINICAL TRIAL: NCT00565786
Title: A Prospective Clinical Data Collection of ArCom® and ArComXL® Polyethylene
Brief Title: ArCom® and ArComXL® Polyethylene Data Collection
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.H011
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ArCom® Polyethylene: ArCom® Polyethylene
  Interventions: Device: ArCom® Polyethylene
- ArComXL® Polyethylene: ArComXL® Polyethylene
  Interventions: Device: ArComXL® Polyethylene

INTERVENTIONS:
Device: ArCom® Polyethylene — Argon packaged compression molded polyethylene
  Groups: ArCom® Polyethylene
Device: ArComXL® Polyethylene — Highly crosslinked Ultra High Molecular Weight Polyethylene
  Groups: ArComXL® Polyethylene

SUMMARY:
The purpose of this prospective clinical data-collection is to document the performance, clinical outcomes, and wear rates of ArCom® and ArComXL® Polyethylene. The data gathered will be collated and used as a part of Biomet's post-market surveillance system and to provide feedback to designing engineers, support marketing efforts, and answer potential questions from reimbursement agencies.

Inclusion/exclusion criteria are identical to those indications and contraindications stated in the FDA approved labeling for the device in 510(k) K926107 and 510(k) K043051. Surgical techniques and patient care are to be standard for the surgeons participating in the protocol.

DETAILED DESCRIPTION:
The study follow-up intervals are 6 weeks, 1 year, 2 years, 3 years, 5 years, and 10 years. Demographic data is collected pre-operatively along with the Harris Hip Score and UCLA Activity Score. Operative information includes the surgical technique and other standard operative information. Follow-up information includes the Harris Hip Score, UCLA Activity Score, and Radiographic data. Anterior/posterior and frog leg lateral X-ray data is recorded to show radiolucencies, component position and angles. Sites are also required to send in an Anterior/Posterior Pelvis x-ray for wear analysis. Implant durability is documented by asking the surgeon to record revisions, complications, and device related adverse events. All information collected is de-identified in compliance with HIPAA regulations.

ELIGIBILITY:
Inclusion Criteria:

* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid arthritis
* Correction of functional deformity
* Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
* Revision of previously failed total hip arthroplasty

Exclusion Criteria:

* Infection
* Sepsis
* Osteomyelitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients requiring total hip replacement.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2004-07; Primary Completion 2017-01-17 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Polyethylene wear rates | 6 weeks, 1 year, 2 year, 3 year, 5 year, and 10 year
  Independent wear analysis of radiographs. The six-week radiographic evaluation will be assessed in comparison to the one-year evaluation in order to determine the early changes of the polyethylene. The difference between the one and two-year evaluations will yield the first true wear rate. We have included a three-year evaluation to reduce the scatter of the linear regression used to calculate the wear rate. The five-year and ten-year evaluations will produce mid and long-term wear rates.

SECONDARY OUTCOMES:
Pain, Function, Absence of Deformity, and Range of Motion | Pre-intervention, 6 weeks, 1 year, 2 year, 3 year, 5 year, and 10 year
  Pain, Function, Absence of Deformity, and Range of Motion will be measured using the Harris Hip Score. On a scale of 0-100, higher scores mean a better outcome.
Physical Activity Level | Surgery, 6 weeks, 1 year, 2 year, 3 year, 5 year, and 10 year
  Physical Activity Level will be measured using the UCLA Activity Scale. On a scale of 1-10, higher scores mean a better outcome.

OTHER OUTCOMES:
Adverse Event | Surgery, 6 weeks, 1 year, 2 year, 3 year, 5 year, and 10 year
  Evaluated by monitoring the frequency and incidence of device related adverse events or unanticipated adverse device effects in investigational subjects.
Survivorship | Surgery, 6 weeks, 1 year, 2 year, 3 year, 5 year, and 10 year
  Analyze survivorship using revision or intended revision as an endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Kacy Arnold, MBA, Study Director — Zimmer Biomet
Locations (3):
- United States (3):
  - Joint Implant Surgeons, Inc., New Albany, Ohio
  - Texas Center for Joint Replacement, Plano, Texas
  - The Kennedy Center for the Hip & Knee, Oshkosh, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided